CLINICAL TRIAL: NCT03867474
Title: Mixed-methods, Feasibility Randomized Control Trial of Mindfulness-Based Stress Reduction (MBSR) With Older Adults Living With Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI): a Primary Care Context
Brief Title: Mindfulness-Based Stress Reduction With Older Adults Living With Cognitive Impairment in Primary Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: Queen's University (Other)
Responsible Party: Principal Investigator, Todd Tran, Principal Investigator, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-0056-E
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-03

CONDITIONS: Feasibility Randomized Control Trial
Keywords: Mindfulness, Primary Care, MBSR, Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: Enrollment, Randomization and Blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (MBSR) (Experimental): Mindfulness-Based Stress Reduction (MBSR) - Intervention Arm
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Control - Usual Care (No Intervention): Control

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — The intervention group will be delivered in a group-based format, for one three-hour session per week for an 8-week period. Each session will consist of mindfulness practice (e.g. lying down body scan, sitting meditation, mindful eating, mindful movements such as walking and light hatha yoga movements) along with an inquiry about the practice. Strategies on stress reactivity, responding to stress, and some basic content on cognitive behaviour therapy principles will also be taught. Participants will be placed in dyads during the group. Homework practice will be given to complete on a daily basis for approximately 30-45 minutes. During week six participants will attend an all-day silent meditation retreat on a Saturday (Total of 10 sessions = 8 sessions, 1 orientation, and 1 all-day retreat).
  Arms: Intervention (MBSR)

SUMMARY:
People living with subjective cognitive decline (SCD) or mild cognitive impairment (MCI) experience less efficiency in performing complex everyday tasks, which may result in a general sense of discontentment and decreased satisfaction with their overall functional performance. Additionally, SCD and MCI have been associated with concomitant anxiety, depressive mood, perceived stress, a decrease in emotional well-being and quality-of-life (QoL) among community-dwelling older adults. These concomitant psychosocial issues may result in emotional distress which further exacerbates cognitive decline.

At the present time, there is a lack of evidence that supports pharmacologic interventions to ameliorate concomitant psychosocial issues with this particular population due to medication side-effects, drug-drug interaction and polypharmacy. Consequently, exploring alternative non-pharmacological interventions to assist in ameliorating psychosocial issues is an important consideration. Secondly, evaluating perceived satisfaction on functional performance with those living with SCD and MCI, and assessing interventions that may support this is also worthwhile to pursue. Primary care providers are often the first point of contact when older adults and their families become concerned about memory problems. Health care professionals, on an interdisciplinary Family Health Team (FHT), such as occupational therapists, are well-positioned to holistically address both the psychosocial and functional needs in a client/family centred way with this growing population in primary care. The study proposes to offer a Mindfulness-Based Stress Reduction (MBSR) program, which is an 8-week program that has been shown to be beneficial in alleviating emotional distress among adults living with physical and psychological issues in the general population.

DETAILED DESCRIPTION:
Purpose: The overarching purpose of this study is to determine whether MBSR is appropriate for a larger clinical trial. AIM 1: To explore the feasibility of conducting a randomized control trial (RCT) of an occupational therapist-led, 8-week MBSR program in an interprofessional primary care setting, with the following objectives: 1a. To assess participant recruitment, intervention adherence, and study retention, 1b. To explore the acceptability of delivering technology-based tablets (iPads) for intervention, and data collection in the MBSR program and 1c. To explore the perspectives of participants and healthcare providers with respect to satisfaction (e.g. the intervention and its delivery), perceived value, barriers to and facilitators of acceptability of this 8-week MBSR program in primary care.

AIM 2: To evaluate the impact of MBSR on satisfaction with functional performance and psychosocial outcomes in individuals with SCD or MCI with the following objectives: 2a. To determine the effect sizes of satisfaction with functional performance and psychosocial outcomes Methods: A convergent mixed-methods, feasibility randomized control trial will be used. Participants will be randomized into an 8-week intervention or control group (usual care) and these groups will be compared at three different time points. Initially, data analysis will involve collecting and analyzing the quantitative and qualitative strands separately. Both qualitative and quantitative data will then be merged for comparative analysis to best understand both the feasibility of a larger clinical trial and to explore preliminary clinical outcomes from the study.

Significance: The results gained from this study will help to determine the feasibility of pursuing a future fully powered trial. Ultimately, this line of research will determine if there are potential benefits of MBSR in improving perceived satisfaction of functional performance and alleviating concomitant psychosocial issues that is associated with those living with SCD and MCI.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* English fluency
* living independently in the community
* self-reported demographic information that includes either the label of SCD or MCI

Exclusion Criteria:

* history of prior participation in any MBSR or other mindfulness-based interventions, or participation in regular (weekly) mindfulness or yoga practice
* low mood as indicated by a 5 or greater on the Geriatric Depression Scale (GDS)
* alcoholism and/or other substance abuse defined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) (American Psychiatric Association, 2013
* Montreal Cognitive Assessment (MoCA) of 23 (+/- 4) or under; and
* if participating in other concurrent group(s) e.g. cognitive behavioural therapy (CBT) or memory training programs in the community, while in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 30 mins
  A client-centred semi-structured interview of client's self-perception of occupational performance issues in the areas of self-care, productivity, and leisure. Five-step process 1. Identification of issues 2. weighting,3. scoring, 4.reassessment and 5. follow-up

SECONDARY OUTCOMES:
Geriatric Anxiety Inventory (GAI) | 10-15 minutes
  The Geriatric Anxiety Inventory (GAI) consists of 20 "Agree/Disagree" items designed to assess typical common anxiety symptoms.
Patient Health Questionnaire-9 (PHQ-9) | 10-15 minutes
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Perceived Stress Scale (PSS) | 10 minutes
  Assessment of global appraisal of stress instead of focusing on a particular event. The focus of the question is reporting on the lives of respondents as i. unpredictable ii. uncontrollable or iii. overloaded. It's a 4-point scale (0-Never and 4-Very Often) with ten questions
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | 5-10 minutes
  A brief measure designed to capture mindfulness in a jargon free and comprehensive way based on Jon Kabat-Zinn's definition of mindfulness.
  The 10-questionnaire has a 4-point scale (1 - rarely and 10-Almost Always).
Quality-of-Life-Alzheimer's Disease (QoL-AD) | 5-10 minutes
  The survey has 13-items covering domains (physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole).
Acceptance and Action Questionnaire (AAQ) | 5-10 minutes
  To measure psychological flexibility and inflexibility.
  Experiential avoidance is significantly associated with a wide array of behavioral problems as well as psychopathology (Wolgast, 2014)

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 10-15 minutes
  A brief cognitive screening tool to detect MCI
Geriatric Depression Scale (GDS) | 10 minutes
  A brief screening instrument for late-life depression

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Womens College Hospital, Family Health Team, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Unsure at the present moment

REFERENCES:
- [Derived] Tran T, Donnelly C, Nalder E, Trothen T, Finlayson M. Mindfulness-based stress reduction for community-dwelling older adults with subjective cognitive decline (SCD) and mild cognitive impairment (MCI) in primary care: a mixed-methods feasibility randomized control trial. BMC Prim Care. 2023 Feb 9;24(1):44. doi: 10.1186/s12875-023-02002-y. PMID 36759766
- [Derived] Tran T, Donnelly C, Nalder EJ, Trothen T, Finlayson M. Occupational therapist-led mindfulness-based stress reduction for older adults living with subjective cognitive decline or mild cognitive impairment in primary care: a feasibility randomised control trial protocol. BMJ Open. 2020 Jun 23;10(6):e035299. doi: 10.1136/bmjopen-2019-035299. PMID 32580984